CLINICAL TRIAL: NCT06107738
Title: IBEX: Phase 2 Trial of Iberdomide + SQ Daratumumab As Post-Autologous Stem Cell Transplant Maintenance Therapy in Multiple Myeloma
Brief Title: Iberdomide and Daratumumab As Maintenance Therapy After an Autologous Stem Cell Transplant for Multiple Myeloma
Acronym: IBEX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Janssen Pharmaceuticals (Industry); Multiple Myeloma Research Consortium (Network)
Responsible Party: Principal Investigator, Jeffrey Zonder, Principal Investigator, Multiple Myeloma Multidisciplinary team leader, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-082; ISR IMO48-025 (Other: Bristol-Myers Squibb); 54767414MMY2092 (Other: Janssen Research and Development LLC); MMRC-095 (Other Grant/Funding Number: Multiple Myeloma Research Consortium (MMRC))
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iberdomide and Daratumumab (Experimental)
  Interventions: Drug: Iberdomide; Drug: Daratumumab/rHuPH20 Co-formulation

INTERVENTIONS:
Drug: Iberdomide — Iberdomide 1.0mg daily for days 1-21 of a 28-day cycle, an increase to 1.3 mg daily on Day 1-21 of a 28-day cycle is allowed at cycle 4 or higher if the 1.0 mg dose was well tolerated.
  Other Names: CC220
Drug: Daratumumab/rHuPH20 Co-formulation — Daratumumab/rHuPH20 will be dosed as follows:
  * Daratumumab/rHuPH20 1800 mg SC days 1, 8, 15, 22 (28-day cycle; cycles 1-2)
  * Daratumumab/rHuPH20 1800 mg SC days 1, 15 (28-day cycle; cycles 3-6)
  * Daratumumab/rHuPH20 1800 mg SC day 1 (28-day cycle; cycles 7-26)
  Other Names: Darzalex FASPRO; Daratumumab and Hyaluronidase-fihj

SUMMARY:
The goal of this phase 2 clinical trial is to learn if patients with Multiple Myeloma who are minimal residual disease positive after initial therapy (including an autologous stem cell transplant [ASCT]) will benefit from maintenance therapy with Iberdomide and subcutaneous (SC) Daratumumab. The main questions it aims to answer are:

* Assess if giving Iberdomide and the SC Daratumumab in the maintenance setting is an effective treatment and warrants further investigation in patients with residual disease
* Is giving Iberdomide and SC Daratumumab maintenance post ASCT a safe option

Participants will:

* provide informed consent and complete screening assessments for eligibility within 28 days of starting treatment
* Screening assessments include specific laboratory tests, a medical history assessment and a physical examination (including temperature, pulse, blood pressure, respirations, height and weight), an assessment of your heart function, a breathing test, cancer imaging, a bone marrow biopsy, minimal residual disease testing (MRD) and a questionnaire
* If eligible, patients will start treatment with Iberdomide (1.0 mg on day 1-21 of each 28 day cycle, with an increase to 1.3 mg on Cycle 4 if the 1.0 mg dose was tolerated, to a maximum of 26 cycles or progressive disease, whichever is first) and SC Daratumumab (1800 mg SC on days 1, 8, 15 and 22 of cycle 1 and 2, then 1800 mg SC on Day 1 and 15 of cycle 3-6 and 1800 mg SC on Day 1 for cycles 7-26 to a maximum of 26 cycles or progressive disease, whichever is first)
* while receiving treatment on study, physical exams (including temperature, pulse, blood pressure, respirations, height and weight), toxicity assessments, laboratory assessments and questionnaires will be done at various times over the course of the 26 cycles
* an MRD assessment is required at 6, 12 and 24 months after starting treatment
* End of treatment will occur once 26 cycles are completed, or cancer has progressed whichever comes first. At that time, specific laboratory tests, a physical examination (including temperature, pulse, blood pressure, respirations, height and weight), cancer imaging, a bone marrow biopsy and minimal residual disease testing (MRD) will occur.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple Myeloma patients who have received prior DARA-containing induction therapy and have attained at least a partial response.
2. Patients who have completed Autologous Stem Cell Transplant (ASCT) 90-150 days prior to registration, without any post-ASCT therapy and without post-ASCT disease progression (according to IMWG criteria)
3. Patients who are Minimal Residual Disease positive (MRD (+)) as measured by the ClonoSEQ assay using a sensitivity of 10-5, measured 90-150 days following ASCT.
4. Prior DARA-containing induction therapy (at least 3 cycles), attaining at least a partial response.
5. Completed ASCT within 90-150 days prior to registration, without any post-ASCT therapy and without evidence of post-ASCT disease progression (according to IMWG criteria)
6. MRD (+) at the time of study enrollment using the clonoSEQ NGS (next-generation sequencing) assay. Patients with an M-spike of ≥ 0.5 g/dL and/or an abnormal free light chain ratio (with an involved serum free light chain of ≥ 10 mg/dL) at enrollment are considered MRD (+) and do not require baseline MRD testing if they have previously had this testing done with successful clonality assessment.
7. ECOG (Eastern Cooperative Oncology Group) Performance Status </= 2
8. Adequate bone marrow function as evidenced by platelets >/= 75,000/mm3, hemoglobin >/= 8 g/dL, and ANC (absolute neutrophil count) >/= 1,000/mm3 within 28 days prior to registration. NOTE: transfusion to achieve the hemoglobin threshold IS permissible.
9. Adequate hepatic function defined by the following within 28 days prior to registration: total bilirubin </=1.5 x IULN (institutional upper limit of the norm, except in case of Gilbert's syndrome) AND AST (aspartate aminotransferase and ALT (aspartate transaminase) </=3.0 x IULN
10. Adequate renal function, as defined by creatinine clearance (CrCl) >/= 30 mL/min., as measured by a 24-hour urine collection or estimated by the Cockcroft and Gault formula within 28 days prior to registration.
11. All ASCT-related toxicities must have recovered to </=Grade 1 (except for alopecia, fatigue and amenorrhea) prior to registration
12. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU (milli-International unit)/mL within 10-14 days prior to registration. FCBP must agree to have a second pregnancy test within 24 hours prior to starting Cycle 1. Further, FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 7 days before starting IBER, during therapy, during dose interruptions and continuing for 28 days following discontinuation of Iberdomide and for 90 days following the discontinuation of daratumumab. FCBP must also agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 28 days after the last dose of iberdomide and for 90 days after the last dose of daratumumab. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy. Females of reproductive potential should be referred to a qualified provider of contraceptive methods, if needed.
13. Men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy, during the study treatment and for 90 days after the last dose of study treatment. They must also agree to not donate sperm during the study and for 90 days after either the last dose of iberdomide or the last dose of daratumumab.
14. Must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
15. Age 18 yrs. old or greater

Exclusion Criteria:

1. Active HIV, or HCV (defined as detectable viremia for any of these conditions).
2. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen[HBsAg]). Patients with resolved infection (i.e., patients who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time PCR (polymerase chain reaction) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded.

   EXCEPTION: Patients with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
3. Unable to assess MRD status at entry or is MRD(-) at 10-5 threshold at entry
4. Heart attack or stroke within 90 days of study enrollment
5. Unable to tolerate required anti-thrombotic or anti-viral prophylaxis
6. Major surgery within 28 days of enrollment
7. Medical, neurologic, or psychiatric condition which renders patient unable to safely comply with study therapy and schedule requirements (including, but not limited to, unstable angina, New York Heart Association Class III-IV congestive heart failure, or uncontrolled cardiac arrhythmia)
8. Intolerance of prior DARA therapy (requiring discontinuation of DARA previously due to toxicity)
9. A history of malignancy (other than multiple myeloma) unless all treatment of that malignancy was completed at least 2 years before consent and the patient has no evidence of disease before the date of enrollment. Exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years.
10. Be exhibiting clinical signs of meningeal or central nervous system involvement due to multiple myeloma.
11. Have known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal.
12. Have known moderate or severe persistent asthma within the past 2 years (see Section 9.2.4), or current uncontrolled asthma of any classification. Note that patients who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study, provided that FEV1 is ≥50% of predicted normal.

    Note: pursuant to exclusion criteria (k) and (l), FEV1 testing is required for patients with suspected COPD or asthma. Patients with FEV1 <50% of predicted normal (or for patients ≥65 years of age, old FEV1 <50% or diffusing capacity of the lung [DLCO] <50%) on screening assessment must be excluded.
13. Have any of the following:

    1. Myocardial infarction within 6 months of enrollment, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV),
    2. Uncontrolled cardiac arrhythmia
14. Have known allergies, hypersensitivity, or intolerance to boron or mannitol, sorbitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to the IB) or known sensitivity to lenalidomide, thalidomide, or pomalidomide.
15. Be pregnant, or breast-feeding, or planning to become pregnant or breast-feed while enrolled in this study or within 90 days after the last dose of study treatment(s). Or, if male, planning to father a child while enrolled in this study or within 90 days after the last dose of study treatment(s).
16. Prolongation of QT interval on screening ECG as defined by a QTc interval > 470 msec using Fridericia's QT correction formula.
17. Use of strong inhibitors or inducers of CYP3A4, P-gp, or BCRP for at least 14 days or 5 half-lives (whichever is shorter) prior to initiating protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD (-) at 12 months | 12 months
  Summarized by a binomial response rate and its associated 2-sided 90% confidence interval (CI) using Pearson-Klopper method.

SECONDARY OUTCOMES:
Rate of Sustained MRD (-) | 24 months
  The rate at which IMWG (International Myeloma Working Group) response category improves by at least one grade during maintenance and the rate of treatment interruptions and dosage adjustments during maintenance will be summarized by a binomial response rate and 2-sided 95% CI using Pearson-Klopper method. Two or more consecutive negative measurements during therapy which are at least 6 months apart.
Progression-Free Survival | 12 months
  Duration from the start date of treatment until the date of progression (as defined by IMWG criteria) or death from any cause.
Progression Free Survival | 24 months
  Duration from the start date of treatment until the date of progression (as defined by IMWG criteria) or death from any cause.
Overall Survival | 12 months
  Duration from the start date of treatment until the date of death from any cause
Overall Survival | 24 months
  Duration from the start date of treatment until the date of death from any cause
Rate on Improvement in IMWG response category | 24 months
  Rate at which IMWG response category improves by at least 1 grade
Frequency of treatment interruptions and dosage adjustments during maintenance | 24 months
  Frequency of treatment interruptions and dosage adjustments during maintenance.
Patient reported Quality of Life (QoL) per EORTC QLQ-C30 | At baseline and day 1 of each treatment cycle until end of treatment
  The 30 question European Organization for Research and Treatment, Quality of Life Questionnaire for cancer patients (EORTC QLQ-C30) is a 30-item subject self-reported questionnaire composed of both multi-item and single scales. The EORTC QLQ-C30 questionnaire is scored using a four-point Likert scale. The scores are then transformed to a scale of 0 to 100, where higher scores indicate better quality of life. The questionnaire includes five functions, nine symptoms, and a global health status.
Patient reported Quality of Life (QoL) per EQ-5D-5L | At baseline and day 1 of each treatment cycle until end of treatment
  The European Organization for Research and Treatment EuroQol (EORTC EQ-5D-5L) questionnaire is a patient reported health-related quality of life questionnaire that consists of two parts: The first part is the EQ-5D descriptive system that measures the respondent's health status in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Items are rated 1=No problem, 2=Slight Problem, 3=Moderate Problem, 4=Severe Problem and 5=Extreme Problem or inability. Part 2 is the EQ visual analogue scale (EQ VAS) records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zonder, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - KCI at McLaren Greater Lansing, Lansing, Michigan

IPD SHARING:
Plan to Share IPD: No